CLINICAL TRIAL: NCT04994405
Title: A Prospective, Double-blinded, Randomized Controlled Trial Evaluating Effectiveness of Lower Tourniquet Pressures in Hand Surgery
Brief Title: Lower Tourniquet Pressure Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-00267
Record Dates: First submitted 2021-07-19; First posted 2021-08-06 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Hand Injuries; Upper Extremity Injury
MeSH Terms: conditions — Hand Injuries; Arm Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Pressure (No Intervention): The extremity tourniquet used during hand surgery for these participants will be the standard pressure of 250 mmHg.
- Lower Tiered Pressures (Experimental): The study intervention is the inflation of the extremity tourniquet to a pressure lower than the standard pressure of 250 mmHg during hand surgery for these participants determined by tiered guidelines based on systolic blood pressure (SBP).
  Interventions: Procedure: Tourniquet Pressure

INTERVENTIONS:
Procedure: Tourniquet Pressure — The procedural intervention will be inflation of a pneumatic tourniquet to a lower than standard pressure as determined by the patient's SBP in hand and upper extremity surgery. The control will be inflation of a pneumatic tourniquet at a standard pressure of 250 mmHg in hand and upper extremity surgery.
  The tourniquet used will be the standard tourniquet used for hand and upper extremity surgery at our institutions - a tourniquet 18 inches in length and 3 inches in width manufactured by Stryker (Kalamazoo, MI) used in conjunction with a protective sleeve matched to the size of the tourniquet cuff which is provided by the manufacturer. Both pieces are supplied in a sterile packaging. No other tourniquets will be used.
  Arms: Lower Tiered Pressures

SUMMARY:
This study design is a prospective, double-blinded, randomized controlled trial evaluating the quality of bloodless surgical field with lower tourniquet pressures based on systolic blood pressure (SBP) compared to standard tourniquet pressures. A secondary goal is to evaluate the effect of lower tourniquet pressures on post-operative tourniquet site pain. The rationale behind the study is to provide evidence-based guidelines on tourniquet use to continue providing quality surgical care while minimizing pain and potential harm to patients.

DETAILED DESCRIPTION:
Patients undergoing hand and upper extremity surgery at our institution will be offered participation in this study. Consenting patients will be randomized in a double-blinded fashion to either standard tourniquet pressure of 250 mmHg or lower tourniquet pressures based on SBP. Demographic data will be recorded as well as details of the surgical procedure. Post-operatively, the operating surgeon will complete a questionnaire about the quality of bloodless surgical field and the patient will complete a questionnaire about post-operative pain. This study will enroll approximately 150 patients. Statistical analysis will be completed to analyze the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient age 18 or older
* Undergoing hand or upper extremity procedure
* Tourniquet is used for procedure
* Willingness and ability to consent

Exclusion Criteria:

* Individuals with procedures that are over 120 minutes in length

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Quality of the bloodless surgical field provided by lower tourniquet pressures | Immediately After surgery in recovery room time
  Surgeon-completed questionnaire rating the quality of the bloodless operative field using a 4-point Likert scale ranging from 1 (excellent) meaning no blood in the surgical field to 4 (poor) meaning blood in the surgical field obscures view throughout the procedure. This survey will be completed immediately post-operatively.

SECONDARY OUTCOMES:
Effect of lower tourniquet pressures based on SBP on post-operative tourniquet site pain | Immediately After surgery in recovery room time
  Patient-completed questionnaire rating their tourniquet site pain post-operatively using the Visual Analogue Scale (VAS) ranging from 0 meaning no pain to 10 meaning worst possible pain. This survey will be completed post-operatively in the recovery unit.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Azad, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - NYU Langone Brooklyn, Brooklyn, New York
  - NYU Langone Orthopedic Hospital, New York, New York
  - NYU Langone Orthopedic Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to ali.azad@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.